CLINICAL TRIAL: NCT00811070
Title: A Phase 1/2 Study Of SKI-606 Administered As A Single Agent In Japanese Subjects With Philadelphia Chromosome Positive Leukemias
Brief Title: Study Evaluating SKI-606 (Bosutinib) In Japanese Subjects With Philadelphia Chromosome Positive Leukemias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A4-2203; B1871007 (Other: Alias Study Number)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: CML. Chronic myelocytic leukemia. Philadelphia Chromosome. Japanese. SKI-606. Bosutinib. Imatinib resistant. Imatinib intolerant
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SKI-606 (Bosutinib)

INTERVENTIONS:
Drug: SKI-606 (Bosutinib) — Formulation: 100 mg Capsule for Part 1, 100 mg tablet for Part1 and Part 2.
  SKI-606 (Bosutinib) will be taken by mouth with water and food as continuous once-daily dosing.

SUMMARY:
This is a two-part safety and efficacy study of SKI-606 in subjects who have Philadelphia chromosome positive leukemias (CML). Part 1 will be a dose-escalation study, in which an escalating dose of SKI-606 (Bosutinib), up to 600 mg, will be studied in subjects with imatinib resistant/refractory or imatinib intolerant chronic phase CML. Part 2 will evaluate the safety and efficacy of the maximum tolerated dose (MTD) of SKI-606 (Bosutinib)identified in Part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Cytogenetic or Polymerase Chain Reaction based diagnosis of Chronic phase of Philadelphia Chromosome Positive Chronic Myelogenous Leukemia:

(Part 1), any phase of Philadelphia Chromosome Positive Chronic Myelogenous Leukemia (Part 2), whose disease is resistant/refractory to full-dose imatinib (400 mg for chronic phase subjects/600 mg for advanced leukemia subjects), or are intolerant of any dose of imatinib.

* Adequate duration of prior imatinib therapy.
* No prior exposure to Src, Abl, or Src/Abl kinase inhibitors other than imatinib.
* Eastern Cooperative Oncology Group Performance Status of 0 or 1 for chronic phase subjects, and 0, 1 or 2 for Advanced Stage subjects.
* At least 7 days since any anti-proliferative treatment (including intrathecal chemotherapy) before the first dose of SKI-606, (except hydroxyurea).
* Recovered to National Cancer Institute grade 0-1, or to baseline, from any toxicities of prior anti-tumor treatment, other than alopecia or thrombocytopenia due to active prior treatment (intolerant subjects).
* At least 3 months post allogeneic stem cell transplantation before the first dose of SKI-606.
* Able to take daily oral capsules reliably.
* Absolute neutrophil count greater than 1,000/mL (Part 1)
* Adequate hepatic, and renal function.
* Documented normal INR if not on oral anticoagulant therapy, or, if on oral anticoagulant therapy consistent target INR less than 3.
* Age should be greater than 20 years and less than 75 years (Part 1), greater than 20 years (Part 2), including women of childbearing potential.
* Willingness of male and female subjects, who are not surgically sterile or postmenopausal, must agree and commit to the use of reliable methods of birth control (oral contraceptives, intrauterine devices, or barrier methods used with a spermicide) for the duration of the study and for 30 days after the last dose of SKI-606.

Exclusion Criteria:

* Subjects with Philadelphia chromosome negative Chronic Myelogenous Leukemia.
* Overt leptomeningeal leukemia. Subjects must be free of CNS involvement according to the symptoms for a minimum of 2 months before the first dose of SKI-606. Subjects with CNS symptoms must have a diagnostic lumbar puncture prior to study enrollment.
* Subjects with extramedullary disease only.
* Ongoing requirement for warfarin or other oral anticoagulant therapy (Part 1).
* Ongoing requirement for hydroxyurea (Part 1).
* Graft Versus Host Disease. a. no previous Graft Versus Host Disease allowed (Part 1). b. no treated or untreated Graft Versus Host Disease within 60 days of first dose (Part 2).
* Major surgery within 14 days or radiotherapy within 7 days before the first dose of SKI-606 (recovery from any previous surgery should be complete before day 1).
* Ongoing clinical requirement for administration of a strong inhibitor or inducer of CYP-3A4 (Part 1).
* History of clinically significant or uncontrolled cardiac disease including: a. history of a clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) b. diagnosed or suspected congenital or acquired prolonged QT syndrome c. history of prolonged QTc d. unexplained syncope e. history of or active congestive heart failure f. myocardial infarction within 12 months. g. Uncontrolled angina or hypertension within 3 months.
* Baseline QTcF greater than 0.45 sec (average of triplicate readings).
* Concomitant use of or need for medications known to prolong the QT interval.
* Uncorrected hypomagnesemia or hypokalemia due to potential effects on the QT interval.
* Recent (within 14 days before the first dose of SKI-606) or ongoing clinically significant gastrointestinal disorder.
* Pregnant or breastfeeding women.
* Evidence of serious active infection, or significant medical or psychiatric illness.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-12; Primary Completion 2013-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (23):
- Japan (23):
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Toyohashi Municipal Hospital, Aichi
  - Japanese Red Cross Nagoya First Hospital, Aichi
  - Aichi Cancer Center, Aichi
  - Akita University Hospital, Akita
  - Chiba University Hospital, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Harasanshin Hospital, Fukuoka
  - Kobe City Medical Center General Hospital, Hyōgo
  - Hospital of Hyogo College of Medicine, Hyōgo
  - Kanazawa University Hospital, Ishikawa
  - Tokai University Hospital, Kanagawa
  - University Hospital,Kyoto Prefectural University of Medicine, Kyoto
  - Okayama University Hospital, Okayama
  - Osaka University Hospital, Osaka
  - Kinki University School of Medicine, Osaka
  - Saga University Hospital, Saga
  - Hamamatsu Medical Univ. HP Faculty of Medicine, Shizuoka
  - Tokyo Metropolitan Cancer&Infectious disease Ctr Komagome Hp, Tokyo
  - Japanese Red Cross Medical Center, Tokyo
  - Jikei University Hospital Daisan, Tokyo

REFERENCES:
- [Derived] Takahashi N, Cortes JE, Sakaida E, Ishizawa K, Ono T, Doki N, Matsumura I, Garcia-Gutierrez V, Rosti G, Ono C, Ohkura M, Tanetsugu Y, Viqueira A, Brummendorf TH. Safety profile of bosutinib in Japanese versus non-Japanese patients with chronic myeloid leukemia: a pooled analysis. Int J Hematol. 2022 Jun;115(6):838-851. doi: 10.1007/s12185-022-03314-y. Epub 2022 Mar 2. PMID 35235189
- [Derived] Takahashi N, Nakaseko C, Kobayashi Y, Miyamura K, Ono C, Koide Y, Fujii Y, Ohnishi K. Long-term treatment with bosutinib in a phase 1/2 study in Japanese chronic myeloid leukemia patients resistant/intolerant to prior tyrosine kinase inhibitor treatment. Int J Hematol. 2017 Sep;106(3):398-410. doi: 10.1007/s12185-017-2239-8. Epub 2017 Apr 13. PMID 28409328
- [Derived] Nakaseko C, Takahashi N, Ishizawa K, Kobayashi Y, Ohashi K, Nakagawa Y, Yamamoto K, Miyamura K, Taniwaki M, Okada M, Kawaguchi T, Shibata A, Fujii Y, Ono C, Ohnishi K. A phase 1/2 study of bosutinib in Japanese adults with Philadelphia chromosome-positive chronic myeloid leukemia. Int J Hematol. 2015 Feb;101(2):154-64. doi: 10.1007/s12185-014-1722-8. Epub 2014 Dec 25. PMID 25540064
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3160A4-2203&StudyName=Study%20Evaluating%20SKI-606%20%28Bosutinib%29%20In%20Japanese%20Subjects%20With%20Philadelphia%20Chromosome%20Positive%20Leukemias

RESULTS

PARTICIPANT FLOW:
Groups:
- Bosutinib Second-line 400 mg (Part 1 ): Single oral dose of bosutinib 400 mg on Day 1 and then bosutinib 400 mg orally once daily was administered continuously from Day 3 in participants with chronic phase second-line imatinib resistant/refractory/intolerant chronic myelogenous leukemia (CML) until disease progression, unacceptable toxicity, or withdrawal of consent occurred. Intra-subject dose escalation up to 600 mg was allowed for lack of efficacy after the safety confirmation of 600 mg cohort.
- Bosutinib Second-line 500 mg (Part 1 ): Single oral dose of bosutinib 500 mg on Day 1 and then bosutinib 500 mg orally once daily was administered continuously from Day 3 in participants with chronic phase second-line imatinib resistant/refractory/intolerant chronic myelogenous leukemia (CML) until disease progression, unacceptable toxicity, or withdrawal of consent occurred. Intra-subject dose escalation up to 600 mg was allowed for lack of efficacy after the safety confirmation of 600 mg cohort.
- Bosutinib Second-line 600 mg (Part 1 ): Single oral dose of bosutinib 600 mg on Day 1 and then bosutinib 600 mg orally once daily was administered continuously from Day 3 in participants with chronic phase second-line imatinib resistant/refractory/intolerant chronic myelogenous leukemia (CML) until disease progression, unacceptable toxicity, or withdrawal of consent occurred.
- Bosutinib Primary Second-line 500 mg (Part 2 ): Bosutinib 500 mg was administered orally once-daily in participants with chronic phase second-line imatinib resistant/refractory/intolerant chronic myelogenous leukemia (CML).Intra-subject dose escalation up to 600 mg was allowed for lack of efficacy.
- Bosutinib Advanced Second-line 500 mg (Part 2 ): Bosutinib 500 mg was administered orally once-daily in participants with accelerated or blast phase second-line imatinib resistant/refractory/intolerant chronic myelogenous leukemia (CML). Intra-subject dose escalation up to 600 mg was allowed for lack of efficacy.
- Bosutinib Exploratory Third-line 500 mg (Part 2 ): Bosutinib 500 mg was administered orally once-daily in participants with chronic or accelerated or blast phase third-line imatinib resistant/refractory/intolerant followed by dasatinib or nilotinib resistant/refractory/intolerant chronic myelogenous leukemia (CML). Intra-subject dose escalation up to 600 mg was allowed for lack of efficacy.
Period: Overall Study
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 ) | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Advanced Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Started | 7 | 7 | 3 | 28 | 7 | 11
Completed | 6 | 6 | 3 | 26 | 2 | 10
Not Completed | 1 | 1 | 0 | 2 | 5 | 1
Not completed — Death | 0 | 0 | 0 | 2 | 5 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 ) | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Advanced Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 ) | Total
Number analyzed (Participants) | 7 | 7 | 3 | 28 | 7 | 11 | 63
Age, Customized [Number; unit: Participants]
  < 65 years | 7 | 4 | 2 | 20 | 3 | 9 | 45
  >= 65 years | 0 | 3 | 1 | 8 | 4 | 2 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 12 | 1 | 4 | 24
  Male | 4 | 5 | 1 | 16 | 6 | 7 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT) - Part 1
Description: DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 clinically-relevant non-hematologic toxicity.
Time Frame: Baseline up to Day 28 (Part 1 )
Population: Participants enrolled in Part 1 of the study were analyzed for DLT. Two participants (1 each in the 400 mg and 500 mg) who discontinued the treatment by Day 28 due to non-safety reasons were excluded from the analysis.
Measure: Number; unit: Participants
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 6 | 6 | 3
Participants | 1 | 1 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) - Part 1
Description: MTD was defined as highest dose level for which no more than 1 participant in a dose cohort experienced DLT.
Time Frame: Baseline up to Day 28 (Part 1 )
Population: as for outcome 1
Measure: Number; unit: mg
Groups:
- All Treated Participants (Part 1 ): All participants who received single oral dose of bosutinib 400 mg, 500 mg or 600 mg on Day 1 and then bosutinib 400 mg, 500 mg or 600 mg orally once daily continuously from Day 3 up to Week 4.
Arm/Group | All Treated Participants (Part 1 )
Number analyzed (Participants) | 15
mg | NA — MTD was not achieved since no more than 1 DLT was observed in any cohort.

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) - Part 1
Time Frame: Before and 1, 2, 3, 4, 6, 8, 24 and 48 hours after administration on Day 1, and before and 1, 2, 3, 4, 6, 8, and 24 hours after administration on Day 15
Population: The pharmacokinetic parameter population was defined as all participants who received at least 1 dose of bosutinib and had at least 1 of the pharmacokinetic parameters of interest.
  n= number of participants analyzed.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 7 | 7 | 3
nanogram per milliliter (ng/mL)
  Day 1 (n = 7, 7, 3) | 131 (29.7) | 128 (23.1) | 155 (44.4)
  Day 15 (n = 5, 4, 2) | 129 (24.4) | 226 (49.5) | 214 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported.

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) - Part 1
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 7 | 7 | 3
hour
  Day 1 (n = 7, 7, 3) | 4.00 [3.97 to 7.90] | 3.95 [3.00 to 5.98] | 3.98 [3.97 to 4.03]
  Day 15 (n = 5, 4, 2) | 4.03 [3.92 to 8.00] | 3.95 [3.93 to 7.98] | 4.00 [3.98 to 4.02]

5. Secondary Outcome: Plasma Decay Half-Life (t1/2) - Part 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Before and 1, 2, 3, 4, 6, 8, 24 and 48 hours after administration on Day 1
Population: The pharmacokinetic parameter population was defined as all participants who received at least 1 dose of bosutinib and had at least 1 of the pharmacokinetic parameters of interest.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 7 | 7 | 3
hour | 16.82 (2.37) | 16.90 (2.47) | 17.27 (3.64)

6. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) - Part 1
Description: Area under the plasma concentration time-curve from zero to infinity. AUC on Day 15 was assessed as the steady state AUC.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng•hr/mL)
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 7 | 7 | 3
nanogram*hour per milliliter (ng•hr/mL)
  Day 1 (n = 7, 7, 3) | 2474 (482.7) | 2720 (560.4) | 2760 (625.9)
  Day 15 (n = 5, 4, 2) | 2235 (220.1) | 3690 (962.1) | 3371 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported.

7. Secondary Outcome: Apparent Oral Clearance (CL/F) - Part 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F on Day 15 was assessed as the steady state CL/F.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 7 | 7 | 3
L/hr
  Day 1 (n = 7, 7, 3) | 167 (34.6) | 190 (37.8) | 224 (45.7)
  Day 15 (n = 5, 4, 2) | 180 (17.4) | 144 (41.8) | 179 (NA) — Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported.

8. Secondary Outcome: Apparent Volume of Distribution (Vz/F) - Part 1
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: Before and 1, 2, 3, 4, 6, 8, 24 and 48 hours after administration on Day 1
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 7 | 7 | 3
liter | 4035 (879.8) | 4570 (713.8) | 5707 (2187)

9. Secondary Outcome: Accumulation Ratio (R) - Part 1
Description: R=accumulation ratio (AUCss on Day 15/AUC[0-24] on Day 1)
Time Frame: as for outcome 3
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 5 | 4 | 2
ratio | 1.67 (0.369) | 2.16 (0.556) | 2.46 (NA) — Standard deviation was Standard deviation obtained by sampling distribution of 2 participants was not meaningful, hence not reported.

10. Primary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR) at Week 24 in Chronic Phase Second-line Cohort - Part 2
Description: Cytogenetic response (CyR) is based on the prevalence of Philadelphia chromosome positive (Ph+) cells. Major cytogenetic response was categorized as either complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). CCyR was achieved when there was 0 percent (%) Ph+ cells and PCyR was achieved when 1 to 35% Ph+ cells.
Time Frame: Week 24
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Primary Second-line 500 mg (Part 2 )
Number analyzed (Participants) | 28
percentage of participants | 35.7 [18.6 to 55.9]

11. Secondary Outcome: Percentage of Participants With Maintained Major Cytogenetic Response (MCyR) at Week 24 in Chronic Phase Second-line and Third-line Cohort - Part 2
Description: Cytogenetic response (CyR) is based on the prevalence of Philadelphia positive (Ph+) cells. Major cytogenetic response was categorized as either complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). CCyR was achieved when there was 0 percent (%) Ph+ cells and PCyR was achieved when 1 to 35% Ph+ cells.
  The responder for maintained MCyR included 'participants without baseline response who had a response at a specified time' and 'participants with baseline response who had a post-baseline response either maintained or improved at a specified time'.
Time Frame: Week 24
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Advanced Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Number analyzed (Participants) | 28 | 7 | 11
percentage of participants | 64.3 [44.1 to 81.4] | 14.3 [0.4 to 57.9] | 63.6 [30.8 to 89.1]

12. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR) at Week 24 - Part 1
Description: Cytogenetic response (CyR) is based on the prevalence of Philadelphia positive (Ph+) cells. Major cytogenetic response was categorized as either complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). CCyR was achieved when there was 0 percent (%) Ph+ cells and PCyR was achieved when 1 to 35% Ph+ cells.
Time Frame: Week 24
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Second-line 400 mg (Part 1 ) | Bosutinib Second-line 500 mg (Part 1 ) | Bosutinib Second-line 600 mg (Part 1 )
Number analyzed (Participants) | 7 | 7 | 3
percentage of participants | 42.9 [9.9 to 81.6] | 57.1 [18.4 to 90.1] | 33.3 [0.8 to 90.6]

13. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR) at Week 24 in Chronic Phase Third-line Cohort - Part 2
Description: as for outcome 12
Time Frame: Week 24
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Number analyzed (Participants) | 11
percentage of participants | 18.2 [2.3 to 51.8]

14. Secondary Outcome: Time to Major Cytogenetic Response (MCyR) in Chronic Phase Second-line and Third-line Cohort - Part 2
Description: Time to MCyR was the interval from the date of first dose of study medication until the first date of achieving a given response.
  Time to response in weeks = (event date minus first dose date plus 1)/7, where the event date is the non-missing date of the first attained response or last cytogenetic assessment date of a participants.
Time Frame: 204 weeks in the second-line participants and 48 weeks in the third-line participants
Population: Subset of participants who had the response among all treated population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Number analyzed (Participants) | 13 | 2
weeks | 12.3 [12.0 to 24.1] | 18.1 [12.1 to 24.1]

15. Secondary Outcome: Duration of Major Cytogenetic Response (MCyR) in Chronic Phase Second-line and Third-line Cohort - Part 2
Description: Duration of MCyR was defined as the interval from the date of the earliest demonstration of a response, until the earliest date of loss of that response. Duration of response in weeks = (date of confirmed loss of first attained response minus date of first attained response)/7 days.
Time Frame: 204 weeks in the second-line participants and 48 weeks in the third-line participants
Population: Subset of participants who had the response among all treated population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Number analyzed (Participants) | 13 | 2
weeks | NA [NA to NA] — Median and 95% CI was not estimable due to the small number of responders who lost the response. | NA [NA to NA] — Median and 95% CI was not estimable due to the small number of responders who lost the response.

16. Secondary Outcome: Percentage of Participants With Complete Hematologic Response (CHR) up to Week 192 in Advance Phase Second-line Cohort - Part 2
Description: CHR response was considered to be achieved if participants met all of the following criteria: White Blood Cells =< institutional upper limit of normal, no peripheral blood blasts or promyelocytes, myelocytes+metamyelocytes <5% in blood, absolute neutrophil count >=1.0*10^9 per liter (/L), platelets >=100 but <450*10^9/L, <20% basophils in blood and no extramedulary involvement (including hepato- or splenomegaly), =<5% BM blasts.
Time Frame: Baseline up to Week 192
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Advanced Second-line 500 mg (Part 2 )
Number analyzed (Participants) | 7
percentage of participants | 14.3 [0.4 to 57.9]

17. Secondary Outcome: Time to Achieve Complete Hematologic Response (CHR) in Advanced Phase Second-line Cohort - Part 2
Description: The time to CHR was measured from the date of first dosing to the first date of response. Time to response in weeks = (event date - first dose date plus 1)/7, where the event date is the non-missing date of the first attained response or last assessment date of a participant.
Time Frame: Baseline up to Week 192
Population: Subset of participants who had the response among all treated population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib Advanced Second-line 500 mg (Part 2 )
Number analyzed (Participants) | 1
weeks | 84.0 [NA to NA] — Only 1 participant was analyzed, therefore, 95% CI was not calculated

18. Secondary Outcome: Duration of Complete Hematologic Response (CHR) in Advanced Phase Second-line Cohort - Part 2
Description: The duration of CHR was defined as the interval from the first date of response until the first date of confirmed loss of response. Duration of response in weeks =(date of confirmed loss of first attained response - date of first attained response)/7.
Time Frame: Baseline up to Week 192
Population: Subset of participants who had the response among all treated population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib Advanced Second-line 500 mg (Part 2 )
Number analyzed (Participants) | 1
weeks | 95.3 [NA to NA] — Only 1 participant was analyzed, therefore, 95% CI was not calculated

19. Secondary Outcome: Percentage of Participants With Overall Hematologic Response (OHR) Up to Week 192 in Accelerated Phase/Blast Phase Third-line Cohort - Part 2
Description: OHR included CHR, no evidence of leukemia (NEL), minor hematologic response (MiHR) or return to chronic phase (RCP), participants had to meet at least 1 of this criterion. Criteria for RCP: disappearance of features defining AP/BP, but still in CP and persistence of clonal evolution. Criteria for MiHR: <15% blasts in blood and bone marrow, <30% blasts+promyelocytes in blood and bone marrow, <20% basophils in blood, no extramedullary disease other than liver/spleen. Criteria for CHR and NEL: <20% basophils in blood, no extramedullary involvement including liver/spleen, no peripheral blasts or promyelocytes, myelocytes + metamyelocytes <5% in blood, <5% (NEL) and <=5% (CHR) marrow blasts, 0.5*10^9 <= Absolute neutrophil count (ANC) <1.0*10^9/L (NEL) and ANC>=1.0*10^9/L (CHR), 20*10^9 <=platelets<100 *10^9/L (NEL) and platelets>=100 but <450x10^9/L (CHR), white blood cells <=institutional upper limit of the normal range.
Time Frame: Baseline up to Week 192
Population: Subset of the third-line cohort who was in accelerated or blast phase
Measure: Number; unit: percentage of participants
Groups:
- Bosutinib Exploratory Third-line 500 mg - AP/BP (Part 2 ): Bosutinib 500 mg was administered orally once-daily in participants with accelerated or blast phase (AP/BP) third-line imatinib resistant/intolerant followed by dasatinib or nilotinib resistant/intolerant chronic myelogenous leukemia (CML). Intra-subject dose escalation up to 600 mg was allowed for lack of efficacy.
Arm/Group | Bosutinib Exploratory Third-line 500 mg - AP/BP (Part 2 )
Number analyzed (Participants) | 1
percentage of participants | 100

20. Secondary Outcome: Time to Achieve Overall Hematologic Response (OHR) in Accelerated Phase/Blast Phase Third-line Cohort - Part 2
Description: The time to OHR was measured from the date of first dosing to the first date of response. Time to response in weeks = (event date - first dose date plus 1)/7, where the event date is the non-missing date of the first attained response or last assessment date of a participant.
Time Frame: Baseline up to Week 192
Population: Subset of participants who had the response among all treated population and who was in accelerated or blast phase in the third-line cohort
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib Exploratory Third-line 500 mg - AP/BP (Part 2 )
Number analyzed (Participants) | 1
weeks | 12.4 [NA to NA] — Only 1 participant was analyzed, therefore, 95% CI was not calculated

21. Secondary Outcome: Duration of Overall Hematologic Response (OHR) in Accelerated Phase/Blast Phase Third-line Cohort - Part 2
Description: The duration of OHR was defined as the interval from the first date of response until the first date of confirmed loss of response. Duration of response in weeks =(date of confirmed loss of first attained response - date of first attained response)/7.
Time Frame: Baseline up to Week 192
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Bosutinib Exploratory Third-line 500 mg - AP/BP (Part 2 )
Number analyzed (Participants) | 1
weeks | 36.1 [NA to NA] — Only 1 participant was analyzed, therefore, 95% CI was not calculated.

22. Secondary Outcome: Time to Treatment Failure (TTF) Rate - Part 2
Description: TTF was the interval from the date of first dose of bosutinib until the earlier date of progression or death (any cause), withdrawal from treatment owing to an AE, subject refusal, or loss to follow-up (censored at the last contact date), or further anti-tumor therapy before documented progression (whichever occurred first). TTF rate indicates the probability of no treatment failure. Percent of participants with no treatment failure were estimated.
Time Frame: Date of first dose of study drug up to Week 336 in primary second line participants; up to Week 192 in advanced second line and exploratory third line participants
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Advanced Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Number analyzed (Participants) | 28 | 7 | 11
percentage of participants
  Week 48 | 67.9 [50.6 to 85.2] | 14.3 [0.0 to 40.2] | 81.8 [59.0 to 100]
  Week 96 | 60.7 [42.6 to 78.8] | 14.3 [0.0 to 40.2] | 72.7 [46.4 to 99.0]
  Week 144 | 57.1 [38.8 to 75.5] | 14.3 [0.0 to 40.2] | 63.6 [35.2 to 92.1]
  Week 192 | 53.6 [35.1 to 72.0] | NA [NA to NA] — TTF rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 179. | NA [NA to NA] — TTF rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 160.
  Week 240 | 53.6 [35.1 to 72.0] | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.
  Week 288 | 45.9 [24.9 to 67.0] | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.
  Week 336 | NA [NA to NA] — TTF rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 312. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.

23. Secondary Outcome: Progression-free Survival (PFS) Rate - Part 2
Description: PFS was based on Kaplan-Meier estimates. PFS was defined as time in weeks from start of study treatment to treatment discontinuation due to disease progression as assessed by the investigator. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from death case report forms (CRFs). Percent of participants with PFS were estimated.
Time Frame: as for outcome 22
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Advanced Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Number analyzed (Participants) | 28 | 7 | 11
percentage of participants
  Week 48 | 100 [100 to 100] | 21.4 [0.0 to 56.3] | 100 [100 to 100]
  Week 96 | 94.4 [83.9 to 100] | 21.4 [0.0 to 56.3] | 88.9 [68.4 to 100]
  Week 144 | 94.4 [83.9 to 100] | 21.4 [0.0 to 56.3] | 88.9 [68.4 to 100]
  Week 192 | 94.4 [83.9 to 100] | NA [NA to NA] — PFS rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 179. | NA [NA to NA] — PFS rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 160.
  Week 240 | 94.4 [83.9 to 100] | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.
  Week 288 | 94.4 [83.9 to 100] | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.
  Week 336 | NA [NA to NA] — PFS rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 312. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.

24. Secondary Outcome: Overall Survival (OS) Rate - Part 2
Description: OS was based on Kaplan-Meier method. Survival was defined as the time period from the date of first dose of bosutinib to the date of death, censored at the participant's last contact date. Percent of participants with OS were estimated.
Time Frame: as for outcome 22
Population: All treated population was defined as all participants who received at least 1 dose of bosutinib.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bosutinib Primary Second-line 500 mg (Part 2 ) | Bosutinib Advanced Second-line 500 mg (Part 2 ) | Bosutinib Exploratory Third-line 500 mg (Part 2 )
Number analyzed (Participants) | 28 | 7 | 11
percentage of participants
  Week 48 | 96.4 [89.6 to 100] | 42.9 [6.2 to 79.5] | 100 [100 to 100]
  Week 96 | 96.4 [89.6 to 100] | 42.9 [6.2 to 79.5] | 100 [100 to 100]
  Week 144 | 96.4 [89.6 to 100] | 28.6 [0.0 to 62.0] | 100 [100 to 100]
  Week 192 | 96.4 [89.6 to 100] | NA [NA to NA] — OS rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 179. | NA [NA to NA] — OS rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 160.
  Week 240 | 96.4 [89.6 to 100] | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.
  Week 288 | 82.7 [57.0 to 100] | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.
  Week 336 | NA [NA to NA] — OS rate and 95% CI was not calculated as all participants were discontinued the follow up by Week 312. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192. | NA [NA to NA] — Data was not collected as participants were only assessed up to Week 192.

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Groups:
- Total Second-line: All participants who received bosutinib orally once daily in second-line chronic myelogenous leukemia (CML), who were imatinib resistant/refractory/intolerant.
- Exploratory Third-line: All participants who received bosutinib 500 mg orally once daily in third-line chronic myelogenous leukemia (CML), participants were with imatinib resistant/refractory/intolerant followed by dasatinib or nilotinib resistant/refractory/intolerant.
- Total Population: Total participants who were second-line or third-line chronic myelogenous leukemia (CML).
Arm/Group | Total Second-line | Exploratory Third-line | Total Population
Serious Adverse Events (participants affected / at risk) | 19/52 | 2/11 | 21/63
Other Adverse Events (participants affected / at risk) | 52/52 | 11/11 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Second-line (N=52) | Exploratory Third-line (N=11) | Total Population (N=63)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 1 | 2
Macular fibrosis (Eye disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Pertussis (Infections and infestations) | 1 | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Macular hole (Eye disorders) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Second-line (N=52) | Exploratory Third-line (N=11) | Total Population (N=63)
Anaemia (Blood and lymphatic system disorders) | 13 | 0 | 13
Eosinophilia (Blood and lymphatic system disorders) | 3 | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 11 | 2 | 13
Lymphopenia (Blood and lymphatic system disorders) | 19 | 5 | 24
Neutropenia (Blood and lymphatic system disorders) | 12 | 2 | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 2 | 18
Conjunctival haemorrhage (Eye disorders) | 3 | 0 | 3
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 7 | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2 | 9
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 7 | 0 | 7
Dental caries (Gastrointestinal disorders) | 9 | 2 | 11
Diarrhoea (Gastrointestinal disorders) | 50 | 10 | 60
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 5
Gastritis (Gastrointestinal disorders) | 7 | 0 | 7
Nausea (Gastrointestinal disorders) | 19 | 5 | 24
Proctalgia (Gastrointestinal disorders) | 4 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 11 | 1 | 12
Vomiting (Gastrointestinal disorders) | 22 | 1 | 23
Chest discomfort (General disorders) | 3 | 0 | 3
Chills (General disorders) | 1 | 1 | 2
Fatigue (General disorders) | 7 | 1 | 8
Malaise (General disorders) | 3 | 1 | 4
Pyrexia (General disorders) | 12 | 0 | 12
Hepatic function abnormal (Hepatobiliary disorders) | 7 | 2 | 9
Liver disorder (Hepatobiliary disorders) | 1 | 1 | 2
Bronchitis (Infections and infestations) | 4 | 0 | 4
Cystitis (Infections and infestations) | 3 | 1 | 4
Folliculitis (Infections and infestations) | 3 | 0 | 3
Gastroenteritis (Infections and infestations) | 8 | 0 | 8
Gingivitis (Infections and infestations) | 6 | 1 | 7
Influenza (Infections and infestations) | 5 | 0 | 5
Nasopharyngitis (Infections and infestations) | 30 | 6 | 36
Otitis media (Infections and infestations) | 0 | 1 | 1
Periodontitis (Infections and infestations) | 3 | 0 | 3
Pharyngitis (Infections and infestations) | 5 | 0 | 5
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1 | 2
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 20 | 4 | 24
Amylase increased (Investigations) | 6 | 1 | 7
Aspartate aminotransferase increased (Investigations) | 15 | 4 | 19
Blood albumin decreased (Investigations) | 4 | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 9 | 2 | 11
Blood bilirubin increased (Investigations) | 1 | 1 | 2
Blood creatine phosphokinase decreased (Investigations) | 3 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 6 | 2 | 8
Blood creatinine increased (Investigations) | 8 | 0 | 8
Blood lactate dehydrogenase increased (Investigations) | 4 | 2 | 6
Blood sodium decreased (Investigations) | 3 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 9 | 1 | 10
Haemoglobin decreased (Investigations) | 6 | 0 | 6
Lipase increased (Investigations) | 11 | 4 | 15
Liver function test abnormal (Investigations) | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 2 | 1 | 3
Platelet count decreased (Investigations) | 3 | 0 | 3
Weight decreased (Investigations) | 9 | 0 | 9
White blood cell count decreased (Investigations) | 3 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 14 | 1 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 4
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 0 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 2 | 1 | 3
Headache (Nervous system disorders) | 4 | 1 | 5
Somnolence (Nervous system disorders) | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 4 | 0 | 4
Renal impairment (Renal and urinary disorders) | 3 | 0 | 3
Urogenital haemorrhage (Renal and urinary disorders) | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 8
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
Acne (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 5
Eczema (Skin and subcutaneous tissue disorders) | 6 | 0 | 6
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Leukoderma (Skin and subcutaneous tissue disorders) | 3 | 0 | 3
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2 | 8
Rash (Skin and subcutaneous tissue disorders) | 31 | 5 | 36
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 5 | 0 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Hypertension (Vascular disorders) | 6 | 0 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 0 | 3
Pericardial effusion (Cardiac disorders) | 4 | 0 | 4
Cataract (Eye disorders) | 3 | 1 | 4
Enterocolitis (Gastrointestinal disorders) | 3 | 0 | 3
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 1
Periodontal disease (Gastrointestinal disorders) | 3 | 0 | 3
Conjunctivitis (Infections and infestations) | 3 | 1 | 4
Epididymitis (Infections and infestations) | 1 | 1 | 2
Herpes zoster (Infections and infestations) | 3 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 0 | 3
Blood potassium increased (Investigations) | 1 | 1 | 2
Blood uric acid increased (Investigations) | 0 | 1 | 1
Weight increased (Investigations) | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Dysgeusia (Nervous system disorders) | 1 | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.